CLINICAL TRIAL: NCT03751644
Title: Peripherical Neuromuscular Electrical Stimulation in Systemic Autoimmune Myopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Samuel Katsuyuki Shinjo, PhD, Professor, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MYO-HCFMUSP-07
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Electrical Remodeling; Rheumatic Diseases; Myopathy
Keywords: systemic autoimmune myopathies; Peripherical neuromuscular electrical stimulation; myositis
MeSH Terms: conditions — Atrial Remodeling; Rheumatic Diseases; Muscular Diseases; Myositis | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with systemic autoimmune myopathies will receive or not the periphericalneuromuscular electrical stimulation in thigh muscles
Who Masked: Investigator
Masking Description: Patients will be randomized by non-investigator from the present study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical stimulation (Experimental): After local antisepsis, 4 electrodes will be placed at the proximal and distal extremities of the lateral and vastus medialis muscles of dominant limb. A positive, single-phase pulsating (intermittent) current with a rectangular waveform will be delivered with a duty cycle of 10 to 15 seconds shutdown at a frequency of 60 Hertz with a pulse width of 400 microseconds for 30 minutes. To control the degree of muscle activation, electrical stimulation will be administered at an intensity that will consistently produce a target torque equal to 15% of maximal voluntary contraction, as monitored in real time through torque output. The desired intensity of stimulation and intensity adjustments throughout the treatment will be evaluated in all patients.
  Interventions: Other: Electrical stimulation
- Placebo (No Intervention): Patients will not submitted to electrical stimulation.

INTERVENTIONS:
Other: Electrical stimulation — Patients with systemic autoimmune myopathies will receive peripheral electrical stimulation in thigh muscles
  Arms: Electrical stimulation

SUMMARY:
Systemic autoimmune myopathies are a heterogeneous group of rheumatic diseases with progressive skeletal muscle weakness. The relevance of the peripherical neuromuscular electrical stimulation has never applied in the patients with systemic autoimmune myopathies. Therefore, the main objective of the present prospective, randomized, investigator-blind, placebo-controlled study is to evaluate the safety and efficacy of the application of an acute peripherical neuromuscular electrical stimulation session in patients with systemic autoimmune myopathies.

DETAILED DESCRIPTION:
Systemic autoimmune myopathies are a heterogeneous group of rheumatic diseases that primarily affect the skeletal muscles. Despite these advances, this group of diseases still continues to be associated with high morbidity and functional disability, mainly due to the proximal muscular weakness of the scapular and pelvic girdles that may prevent the total recovery of these patients. On the other hand, the importance of the peripherical neuromuscular electrical stimulation has never applied in the patients with systemic autoimmune myopathies. Therefore, the main objective of the present prospective, randomized, investigator-blind, placebo-controlled study is to evaluate the safety and efficacy of the application of an acute peripherical neuromuscular electrical stimulation session in patients with systemic autoimmune myopathies.

ELIGIBILITY:
Inclusion Criteria:

* Classification criteria - EULAR/ACR 2017
* Classification criteria - Connors et al.
* Objective muscle limb weakness

Exclusion Criteria:

* Neoplasia
* Using heart pacemarker
* Using visceral metalic clips
* Infections (HIV, HTLV-1, Hepatitis, etc)
* Pregnancy
* Previous historical of convulsions or epilepsies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 6 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events [safety and tolerability] | 30 minutes after stimulation
  Frequency of disease relapsing (based on the questionnaire of secondary outcome measures) and tolerability (patients' symptom registration) electrical stimulation in patients with systemic autoimmune myopathies.
Frequency of treatment-emergent adverse events [safety and tolerability] | 8 weeks after stimulation
  Frequency of disease relapsing (based on the questionnaire of secondary outcome

SECONDARY OUTCOMES:
Healthy Assessment Questionnaire (HAQ) | 3 times: (a) within 30 minutes before stimulation. Then, after (b) 3 weeks and (c) 8 weeks after stimulation
  Specific questionnaires to assess the quality of life. Pontuaction: 0.00 (best) - 3.00 (worst)
Patient/Parent Global Activity | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale. Pontuaction: 0 (best) - 10 (worst)
Physician Global Activity | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. Pontuaction: 0 (best) - 10 (worst)
Manual Muscle Testing | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies. Pontuaction 0 (worst) - 80 (best)
Myositis Disease Activity Assessment Visual Analogue Scales (MYOACT) | 3 times: (a) within 30 minutes before stimulation. Then, after (b) 3 weeks and (c) 8 weeks after stimulation
  This partially validated tool measures the degree of disease activity of extra-muscular organ systems and muscle. The questionnaire is a series of physician's assessments of disease activity. Score ranges: 0 (best) - 60 (worst).
Serum levels of muscle enzymes | 4 times: (a) within 30 min before; (b) until 30 min after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  This partially validated tool measures the serum activities of at least 2 of the 4 muscle-associated enzymes including creatine phosphokinase (CK), the transaminases (ALT, AST), lactate dehydrogenase (LD) and aldolase. International Unit: U/L.
Strength muscle tests | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  The dynamic 1-repetition maximum for the leg-press will be assessed at baseline and after the intervention. Strength unit: Newton (N). The values vary according to each patient.
Strength muscle tests | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  The dynamic 1-repetition maximum for the bench-press exercises will be assessed at baseline and after the intervention. Strength unit: Newton (N). The values vary according to each patient.
Strength muscle tests | 4 times: (a) within 30 minutes before; (b) until 30 minutes after stimulation. Then, after (c) 3 weeks and (d) 8 weeks after stimulation
  Isometric strength (assessed by handgrip, with the dominant arm) will be assessed at baseline and after the intervention. Strength unit: Newton (N). The values vary according to each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel K Shinjo, Principal Investigator — Universidade de Sao Paulo - Rheumatology Division
Locations (1):
- Samuel K Shinjo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided